CLINICAL TRIAL: NCT00452868
Title: A Pilot Study of Donepezil Hydrochloride in Pediatric Brain Tumor Survivors After Cranial Irradiation
Brief Title: Donepezil in Treating Young Patients With Primary Brain Tumors Previously Treated With Radiation Therapy to the Brain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000537049; P30CA012197 (NIH); CCCWFU-91305 (Other: Comprehensive Cancer Center of WFUHS); CCCWFU-IRB-00000258 (Other: WFUHS IRB)
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Long-term Effects Secondary to Cancer Therapy in Children; Neurotoxicity; Psychosocial Effects of Cancer and Its Treatment; Radiation Toxicity
Keywords: cognitive/functional effects; neurotoxicity; long-term effects secondary to cancer therapy in children; psychosocial effects of cancer and its treatment; radiation toxicity; childhood central nervous system germ cell tumor; childhood choroid plexus tumor; childhood craniopharyngioma; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; childhood spinal cord neoplasm; childhood brain stem glioma; childhood cerebellar astrocytoma; childhood medulloblastoma; childhood supratentorial primitive neuroectodermal tumor; childhood visual pathway and hypothalamic glioma; childhood subependymal giant cell astrocytoma; childhood ependymoma; childhood cerebral astrocytoma/malignant glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neurotoxicity Syndromes; Radiation Injuries; Choroid Plexus Neoplasms; Spinal Cord Neoplasms; Medulloblastoma; Optic Nerve Glioma; Astrocytoma; Familial ependymoma | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Donepozil (Experimental): Donepezil 5 milligrams a day for 6 weeks
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Donepezil 5 milligrams a day for 6 weeks

SUMMARY:
RATIONALE: Donepezil may decrease the side effects caused by radiation therapy to the brain.

PURPOSE: This clinical trial is studying how well donepezil works in treating young patients with primary brain tumors previously treated with radiation therapy to the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the impact of donepezil hydrochloride on cognitive function in pediatric patients with primary brain tumors previously treated with cranial radiotherapy.

Secondary

* Assess health-related quality of life of patients treated with this drug.
* Assess function and quality of life of the families of patients treated with this drug.
* Determine the physiologic effects of radiotherapy on cerebrovascular hemodynamics in patients treated with this drug.
* Determine the toxicity of donepezil hydrochloride in these patients.

OUTLINE: This is a multicenter, pilot, open-label, controlled study.

Patients receive oral donepezil hydrochloride once daily or once every other day for up to 24 weeks in the absence of disease progression or unacceptable toxicity. After completion of 6 weeks of study therapy, patients are evaluated for toxicity. Patients experiencing no adverse effects from treatment may continue receiving donepezil hydrochloride at a higher dose for 18 more weeks.

Patients undergo measurement of cognitive function (by neurocognitive testing), behavioral adjustment and social competency (by parent-reported questionnaires), health-related quality of life (by child- and parent-reported questionnaires), and vascular dynamics (by transcranial Doppler ultrasound) at baseline and at weeks 12, 24, and 36. Family function and family quality of life are assessed at baseline and at week 24.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of primary brain tumor
* No type 2 neurofibromatosis
* Underwent fractionated radiotherapy (≥ 23.4 Gy) with or without surgery or chemotherapy for the brain tumor at least 1 year ago
* Karnofsky or Lansky performance status 70-100%
* Fertile patients willing to use effective contraception
* Baseline IQ ≥ 70 on Peabody Picture Vocabulary Test-3
* Stable weight within the past 6 months with no concern of weight loss
* Vision aids and hearing aids must be used for all neuropsychologic/neurocognitive tests, If indicated
* Able to speak English
* More than 6 weeks since prior donepezil hydrochloride, EGb761, methylphenidate hydrochloride, other stimulants, or any other cognitive function-enhancing drug

Exclusion Criteria:

* Stereotactic radiosurgery as sole treatment
* Evidence of disease progression by MRI
* Pregnant or nursing
* Attention-deficit/hyperactivity disorder before cancer diagnosis
* Uncontrolled seizures or uncontrolled endocrinopathies
* Uncontrolled comorbidities
* Steroid dose greater than physiologic replacement (18-30 mg/m² hydrocortisone or equivalent)
* Use of concurrent anticholinergic drugs

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M. Castellino, MD, FAAP, Study Chair — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were registered from 9/11/2006 to 5/14/2009
Pre-assignment Details: 13 unique patients were recruited, one patient twice after failing to start therapy the first time, two patients were not evaluable, leaving 11 patients for analysis.
Groups:
- Donepezil: Patients less than 35 kilograms(kg): Donepezil 5 milligrams (mg) orally once every alternate day. Patients greater than 35 kg Donepezil 5 mg orally once per day. If there are no adverse effects noted on review of symptoms, the dose will be increased to 5 mg daily for patients < 35 kg. And to 10 mg/day for patients > 35 kg. This evaluation and dose escalation may be done as early as week 4. For all, donepezil will be administered 24 weeks.
Period: Overall Study
Arm/Group | Donepezil
Started | 13
Completed | 11
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Donepezil
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.81 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Neurocognitive Function as Measured by the Neurocognitive Battery at 24 Weeks
Description: Delis-Kaplan Executive Function System Tower Total Scaled Score, range is 1-19 with the higher score being a better outcome.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 11
units on a scale | 10 (3)

ADVERSE EVENTS:
Arm/Group | Donepezil
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=11)
vomiting (Gastrointestinal disorders) | 2 (2)
Dehydration (General disorders) | 1 (1)
ataxia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Donepezil
Nausea (Gastrointestinal disorders) | 6/11 (6)
Diarrhea (Gastrointestinal disorders) | 5/11 (5)
Anorexia (General disorders) | 5/11 (5)
Incontinence, urinary (Renal and urinary disorders) | 1/11 (1)
Personality/behavioral (Psychiatric disorders) | 1/11 (1)
Dizziness (Ear and labyrinth disorders) | 1/11 (1)
Insomnia (Psychiatric disorders) | 4/11 (4)
Neurology (Nervous system disorders) | 2/11 (2)
Fatigue (General disorders) | 10/11 (10)
Pain: Head/headache (Nervous system disorders) | 1/11 (1)
Occular/Visual (Eye disorders) | 2/11 (2)
Fever (in the absence of neutropenia) (Infections and infestations) | 1/11 (1)
Infection (Infections and infestations) | 1/11 (1)
Speech Impairment (Psychiatric disorders) | 1/11 (1)
Confusion (Nervous system disorders) | 1/11 (1)
Mood Alteration: Agitation (Psychiatric disorders) | 1/11 (1)
Pain: Abdomen NOS (General disorders) | 4/11 (4)
Pain: Back (General disorders) | 1/11 (1)
Hemorrhag, pulmonary/upper respiratory: nose (Vascular disorders) | 1/11 (1)
Extrapyramidal/involuntary movement/restlessness (Psychiatric disorders) | 1/11 (1)
Incontenence, anal (Gastrointestinal disorders) | 1/11 (1)
Muscle weakness, generalized: whole body (Musculoskeletal and connective tissue disorders) | 1/11 (1)
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 5/11 (5)
Pain: Extremity-limb (General disorders) | 1/11 (1)
Pain: Skin (Skin and subcutaneous tissue disorders) | 1/11 (1)
Infection with unknown ANC: Bronchus (Infections and infestations) | 1/11 (1)
Infection with unknown ANC: Nerv-peripheral (Infections and infestations) | 1/11 (1)
Infection with unknown ANC: Urinary tract NOS (Infections and infestations) | 1/11 (1)
Muscle weakness, generalid or specfic ara (not due to neuropathy): Left sided (Musculoskeletal and connective tissue disorders) | 1/11 (1)
Neuropathy: cranial: CN VIII Hearing and balance (Ear and labyrinth disorders) | 1/11 (1)

LIMITATIONS AND CAVEATS:
small number (11) analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes